CLINICAL TRIAL: NCT03824301
Title: Comparative Study Between Different Modes of Ventilation During Cardiopulmonary Bypass and Its Effect on Postoperative Pulmonary Dysfunction
Brief Title: Different Modes of Ventilation During Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ayman Anis Metry, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ASCSH32/17
Record Dates: First submitted 2019-01-23; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Pulmonary Dysfunction
Keywords: cardiopulmonary bypass; pressure-controlled ventilation; volume-controlled ventilation; atelectasis; pleural effusion; lung compliance
MeSH Terms: conditions — Pulmonary Atelectasis; Pleural Effusion

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Volume-controlled ventilation (Active Comparator): During cardiopulmonary bypass period the patients were ventilated with volume-controlled ventilation
  Interventions: Device: Volume controlled ventilation
- Pressure-controlled ventilation (Active Comparator): During cardiopulmonary bypass period the patients were ventilated with pressure-controlled ventilation
  Interventions: Device: Pressure controlled ventilation
- No ventilation (No Intervention): During cardiopulmonary bypass period the patients were disconnected from ventilator

INTERVENTIONS:
Device: Volume controlled ventilation — Changing modes of ventilation during cardiopulmonary bypass
  Arms: Volume-controlled ventilation
Device: Pressure controlled ventilation — Applying pressure controlled ventilation during cardiopulmonary bypass Period
  Arms: Pressure-controlled ventilation

SUMMARY:
66 patients divided into 3 groups with different modes of ventilation.

DETAILED DESCRIPTION:
Sixty-six patients going through open-heart surgeries were included in the study, divided into 3 groups (P: pressure controlled ventilation, V: volume controlled ventilation, C: control) in accordance with the mode of ventilation. Patients studied for chest x-ray, lung ultrasound, arterial oxygen partial pressure to fractional inspired oxygen ratio (PaO2/FiO2), Alveolar-arterial oxygen gradient, static lung compliance and dynamic lung compliance, taken after induction of anesthesia, 1h post cardiopulmonary bypass, 1h after arrival to cardiac surgical unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoingvalve surgeries
* Patients undergoing coronary artery bypass grafting surgeries

Exclusion Criteria:

* Emergency cases.
* Off-pump surgeries.
* Patients with chronic lung diseases with forced expiratory volume in first second (FEV1) or forced vital capacity (FVC) less than 40% of the predicted value.
* Massive blood transfusion during surgery.
* Complicated surgeries.
* Redo surgeries.
* Patients with decompensated heart failure prior to surgery.
* Patients refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-01-22 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
chest x-ray | after induction of anesthesia, 1hour post cardiopulmonary bypass and 1hour after arrival to cardiac surgical unit.
  Chest x ray to detect any lung pathology or changes from baseline like pleural effusion, pulmonary edema or pneumonia
lung ultrasonography | after induction of anesthesia, 1hour post cardiopulmonary bypass and 1hour after arrival to cardiac surgical unit.
  Lung ultrasonography to detect any lung changes from baseline or development of consolidation, pulmonary edema or pleural effusion

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University cardiothoracic hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No